CLINICAL TRIAL: NCT06995898
Title: The Vanguard Study: Testing a New Way to Screen for Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NCI-2024-10793; NCI-2024-10793 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CSRN1 (Other: Fred Hutchinson Cancer Center); CSRN1 (Other: DCP); CSRN1 (Other: CTEP); P30CA015704 (NIH); UG1CA286954 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-05-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Bladder Carcinoma; Breast Carcinoma; Colorectal Carcinoma; Esophageal Carcinoma; Gastric Carcinoma; Liver Carcinoma; Lung Carcinoma; Malignant Solid Neoplasm; Ovarian Carcinoma; Pancreatic Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Who Masked: Participant
Masking Description: Four ACCESS Hubs will institute participant blinding to their randomly assigned group. Participants recruited in the remaining ACCESS Hubs will be told the arm to which they have been assigned. The purpose of having some Hubs institute blinding and others unblinded is to assess the impact of blinding on recruitment, participation in standard of care cancer screening, and adherence to the study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm I (Shield MCD test) (Experimental): Participants undergo blood collection for Shield MCD testing at enrollment and after one year on study. Participants at unblinded sites are provided results of tests and those with abnormal results follow up with their clinician for additional testing. Participants at blinded sites are provided abnormal results and will follow up with their clinician for additional testing.
  Interventions: Procedure: Biospecimen Collection; Device: Device Usage; Other: Electronic Health Record Review; Procedure: Multi-Cancer Detection Test; Other: Questionnaire Administration
- Arm II (Avantect MCD test) (Experimental): Participants undergo blood collection for Avantect MCD testing at enrollment and after one year on study. Participants at unblinded sites are provided results of tests and those with abnormal results follow up with their clinician for additional testing. Participants at blinded sites are provided abnormal results and will follow up with their clinician for additional testing.
  Interventions: Procedure: Biospecimen Collection; Device: Device Usage; Other: Electronic Health Record Review; Procedure: Multi-Cancer Detection Test; Other: Questionnaire Administration
- Arm III (Control) (Active Comparator): Participants undergo blood collection at enrollment and after one year on study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Device: Device Usage — Evaluation of MCD tests
  Other Names: Usage of Device
  Arms: Arm I (Shield MCD test); Arm II (Avantect MCD test)
Other: Electronic Health Record Review — Obtain health data
Procedure: Multi-Cancer Detection Test — Undergo Shield MCD test
  Other Names: MCD Assay; MCD Test; MCED Assay; MCED Test; Multi Cancer Detection Assay; Multi Cancer Detection Test; Multi Cancer Early Detection Assay; Multi Cancer Early Detection Test; Multi-Cancer Detection Assay; Multi-Cancer Early Detection Assay; Multi-Cancer Early Detection Test
  Arms: Arm I (Shield MCD test)
Procedure: Multi-Cancer Detection Test — Undergo Avantect MCD test
  Other Names: MCD Assay; MCD Test; MCED Assay; MCED Test; Multi Cancer Detection Assay; Multi Cancer Detection Test; Multi Cancer Early Detection Assay; Multi Cancer Early Detection Test; Multi-Cancer Detection Assay; Multi-Cancer Early Detection Assay; Multi-Cancer Early Detection Test
  Arms: Arm II (Avantect MCD test)
Other: Questionnaire Administration — Study specific questionnaires

SUMMARY:
The Vanguard Study is a feasibility study to explore several aspects of evaluating multi-cancer detection (MCD) tests in a future definitive randomized controlled trial. An MCD test measures markers in the blood in order to screen for multiple cancers simultaneously. There is a need to understand how MCDs may work as cancer screening tools. The goal of cancer screening is to reduce the burden of cancer by identifying cancers before they show symptoms or signs, when treatment is likely to be most effective. In this study, adults aged 45-75 without cancer will be randomly assigned to one of 3 groups: 2 separate MCD test groups or a control group. These two MCD tests will not be compared to each other but will be compared to cancers detected in the control group. This study will provide early information on how well MCD tests perform as cancer screening tools. It will also help researchers understand how patients and their doctors make decisions about their care when the MCD test result comes back as normal (negative) or abnormal (positive).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of recruitment and adherence to protocol-required baseline and follow-up data and blood collection.

II. Assess the feasibility of achieving representative enrollment across participating recruitment sites.

SECONDARY OBJECTIVES:

I. To assess the impact of participant blinding on willingness to participate, adherence to protocol required baseline and follow-up data, blood collection, and rates of standard of care screening.

II. To determine the timeliness of returning test results to participants. III. To understand the factors contributing to lack of diagnostic resolution of an abnormal MCD test.

IV. To examine the effects of participant characteristics, including cancer risk factors and social determinants of health, on all aspects of feasibility.

V. To estimate the proportion of participants receiving an MCD test outside of the trial.

VI. To assess the feasibility of a staggered introduction of the second MCD assay intervention arm.

VII. To estimate the proportion of abnormal MCD tests that are diagnostically resolved, and the time to resolution.

VIII. To compare the proportion of participants who receive standard of care screening during follow-up between the intervention and control arms.

IX. To assess the accuracy of tissue of origin prediction for each MCD assay. X. To estimate the incidence of complications related to diagnostic evaluation of an abnormal MCD test result.

XI. To assess the effect of an abnormal MCD test and diagnostic workup on anxiety and cancer worry.

XII. To evaluate the clinical diagnostic performance of the MCD assays.

EXPLORATORY OBJECTIVES:

I. To estimate rates of late-stage cancer, and the distribution of cancer stage.

II. To estimate assay-targeted cancer-specific mortality of each MCD assay, all cancer-specific mortality, and all-cause mortality.

OUTLINE: Participants are randomized to 1 of 3 arms.

ARM I: Participants undergo blood collection for Shield MCD testing at enrollment and after one year on study. Participants at unblinded sites are provided results of tests and those with abnormal results follow up with their clinician for additional testing. Participants at blinded sites are provided abnormal results and will follow up with their clinician for additional testing.

ARM II: Participants undergo blood collection for Avantect MCD testing at enrollment and after one year on study. Participants at unblinded sites are provided results of tests and those with abnormal results follow up with their clinician for additional testing. Participants at blinded sites are provided abnormal results and will follow up with their clinician for additional testing.

ARM III (Control): Participants undergo blood collection at enrollment and after one year on study.

After completion of study intervention, participants are followed passively up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Ages 45-75 years old
* Agree to provide blood samples for possible MCD testing at enrollment and at 1 year following enrollment
* Agree to allow collection of information from their medical records for study-related purposes
* Understand and be able to complete informed consent and participant questionnaires in English, Spanish, or Arabic

  * Note: Eligibility for Spanish and Arabic languages are at the Hub's discretion

Exclusion Criteria:

* Solid malignant tumor or blood cancer diagnosis, with or without treatment, within the last 5 years

  * Note: Persons with a history of in situ cancers (e.g., ductal carcinoma in situ of the breast, cervical cancer in situ, atypical melanocytic hyperplasia or melanoma in situ) or nonmelanoma skin cancer are eligible
* Ongoing cancer diagnostic work-up
* Ongoing participation in another study of an investigational cancer screening test or technology
* Currently breastfeeding or pregnant, or planning to become pregnant in the next year

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24000 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment onto study | At time of randomization
  The number of participants enrolled into the study compared to trial goals.
Proportion of participants who complete baseline and follow-up questionnaires within 60 days of receipt | Up to 3 years
  The proportion of participants who are complete questionnaires and timing of completion.
Proportion of participants who provide the required blood sample for year 1 for Multi-Cancer Detection (MCD) testing within 90 days of recommended time point | Up to 2 years
  The proportion of participants who have a second blood draw and the timing of the blood draw.
Proportion of participants considered lost to follow-up within 2 years of randomization | Up to 2 years
  The proportion of participants who do not complete study procedures and are not able to be contacted.
Representative enrollment | Up to 2 years
  Meeting or exceeding the trial enrollment goals on a population basis.
Staggered start of intervention arm 2 | Up to 1 year
  Advantages and challenges arising from trial activation with one intervention arm and later addition of a second intervention arm.

SECONDARY OUTCOMES:
Impact of participant blinding | Up to 2 years
  Comparisons between blinded and unblinded sites on participation rates, adherence to protocol-required questionnaires and blood collection, and participation in standard of care screening.
Timely return of MCD test result | Up to 2 years
  The time from receipt of the MCD test result at the Statistics and Data Management Center to the time of receipt of the MCD test result at the ACCESS Hub. The time from receipt of MCD test result at the ACCESS Hub to the time of participant receipt of the MCD test result.
Factors contributing to lack of diagnostic resolution of an abnormal MCD test | Up to 2 years
  Factors that contribute to the inability to determine if a participant has a cancer or rule out cancer.
Contamination | Up to 3 years
  Estimated as the number of participants receiving MCD testing outside the trial.
Effects of participant characteristics | Up to 2 years
  Feasibility outcomes will be reported by participant demographics and cancer risk factors.
Diagnostic resolution following an abnormal MCD test result | Within 12 months following an abnormal MCD test result
  The proportion of participants with a "cancer diagnosis" or "no cancer diagnosis" among all participants with an abnormal MCD test result
Time to diagnostic resolution | Up to 2 years
  The number of days from date of ACCESS Hub receipt of abnormal MCD test result to date of provider-reported diagnostic resolution.
Participation in standard of care screening | Up to 2 years
  The proportion of participants that receive standard of care cancer screening in each arm.
Accuracy of tissue of origin prediction | Up to 2 years
  The proportion of diagnosed cancers that match the tissue of origin predicted by an abnormal (positive) MCD test, for each screening episode.
Complications related to diagnostic evaluation of an abnormal MCD test result | Up to 1 year
  Adverse events occurring in participants undergoing a diagnostic workup following receipt of an abnormal MCD test result.
Anxiety and Cancer Worry Questionnaire | Up to 2 years
  Participant anxiety will be assessed with the Patient Reported Outcomes Measurement Information System instrument. Cancer-related worry will be assessed using the Lehrman Cancer Worry Scale.
Sensitivity of clinical diagnostic performance of each MCD assay | Up to 2 years
  Sensitivity will be estimated for each MCD assay. These sensitivities will also be calculated by early- versus late-stage, and for MCD test-targeted cancers and all cancers.
Specificity of each MCD assay | 1 year
  Specificity will be estimated for each MCD assay.
Test positive rates | Up to 2 years
  The proportion of abnormal MCD tests at each screening episode, and the proportion of participants with at least one abnormal test.
False positives | Up to 2 years
  The number of participants with an abnormal MCD test and no cancer diagnosis.
(Targeted cancer) Positive predictive value (PPV) | Up to 2 years
  The proportion of abnormal MCD tests that result in diagnosis of one of the MCD test-targeted cancers among participants with at least one abnormal test, for each screening episode.
(All cancer) PPV | Up to 2 years
  The proportion of abnormal MCD tests that result in diagnosis of any cancer among participants with at least one abnormal test, for each screening episode.
Interval cancers | 1 year
  The number of MCD test-targeted cancer cases diagnosed within 12 months of a normal MCD test result among participants who received an MCD test, for each screening episode.
Detected cancers | 1 year
  The number of cancer cases diagnosed within a 12-month follow-up period of an abnormal test result among participants who received an MCD test, for each screening episode.
(Targeted cancer) Negative predictive value | 1 year
  The proportion of normal MCD tests that did not result in diagnosis of one of the MCD test-targeted cancers among participants with a normal test, for each screening episode.

OTHER OUTCOMES:
Cancer stage | Up to 12 years
  The stage that a cancer was diagnosed (Surveillance, Epidemiology, and End Results [SEER]).
Early and late stages cancer diagnosis | Up to 12 years
  Counts of early and late-stage cancers by arm, separately for each cancer type. Early stage is defined as in situ or localized (SEER). Late stage is defined as regional or distant stage (SEER).
Targeted cancer-specific mortality of each MCD assay | Up to 12 years
  The fraction of MCD-targeted cancers diagnosed during trial participation that resulted in death.
Cancer-specific mortality | Up to 12 years
  The fraction of all cancers diagnosed during trial participation that resulted in death.
All-cause mortality | Up to 12 years
  The probability of participant death by any cause during trial participation, by arm.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Ramsey, Principal Investigator — Fred Hutchinson Cancer Center
Locations (36):
- United States (36):
  - Kaiser Permanente-Division of Research, Pleasanton, California
  - Keefe Memorial Hospital, Cheyenne Wells, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Health Center - Brownstown, Brownstown, Michigan
  - Henry Ford Health Center - Chesterfield, Chesterfield, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center - Detroit Northwest, Detroit, Michigan
  - Henry Ford Medical Center-Cottage, Grosse Pointe Farms, Michigan
  - Henry Ford Medical Center - Livonia, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford Medical Center - Plymouth, Plymouth, Michigan
  - Henry Ford Medical Center - Royal Oak, Royal Oak, Michigan
  - Henry Ford Medical Center, Sterling Heights, Michigan
  - Henry Ford Medical Center - Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm